CLINICAL TRIAL: NCT01418755
Title: Platelet-rich Plasma in Patients With Tibiofemoral Cartilage Degeneration
Brief Title: Study of Platelet-rich Plasma in Treating Patients With Tibiofemoral Cartilage Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Komzak Martin, M.D. (Other)
Responsible Party: Sponsor-Investigator, Komzak Martin, M.D., Hart Radek, M.D., Ph.D., FRS, prof.; Orthopaedic- Traumatologic department, Hospital Znojmo
Organization: Hospital Znojmo (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT12057
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Cartilage Degeneration
Keywords: Platelet-Rich Plasma; Knee; Tibiofemoral Chondromalacia; Injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- platelet rich plasma injection (Experimental): Fifty consecutive and strictly selected patients, affected by Grade II or III chondromalacia, underwent one year treatment (9 injections) with autologous PRP in a liquid form with 2,0 to 2,5-fold platelets concentration. Outcome measures included the Lysholm, Tegner, IKDC, and Cincinnati scores. Magnetic resonance imaging was used to evaluate cartilage thickness and degree of degeneration.
  Interventions: Biological: platelet rich plasma injection

INTERVENTIONS:
Biological: platelet rich plasma injection — The approximate 2.0 to 2.5-fold platelet concentration (taking into consideration the mean human blood platelet count of 200 000 /μl) was achieved in all specimens. Mean platelet concentration in PRP was 459 000 /μl (range, 407 000 /μl to 513 000 /μl).

SUMMARY:
Recently an articular cartilage repair has been given much attention in the orthopaedic field. Cartilage regeneration capacity is very limited. Optimal approach seems to be a delivery of natural growth factors. Autologous platelet-rich plasma (PRP) contains proliferative and chemoattractant growth factors. The objective of the present study was to determine if PRP can increase tibiofemoral cartilage regeneration and improve knee function.

DETAILED DESCRIPTION:
Fifty consecutive and strictly selected patients, affected by Grade II or III chondromalacia, underwent one year treatment (9 injections) with autologous PRP in a liquid form with 2,0 to 2,5-fold platelets concentration. Outcome measures included hte Lysholm, Tegner, IKDC, and Cincinnati scores. Magnetic resonance imaging was used to evaluate cartilage thickness and degree of degeneration.

ELIGIBILITY:
Inclusion Criteria:

* isolated Grade II or Grade III nontraumatic chondromalacia according to Outerbridge grading scale

Exclusion Criteria:

* Grade I (only softening) or Grade IV (exposed subchondral bone) tibiofemoral chondromalacia;
* patellofemoral chondral damage;
* associated intraarticular lesions confirmed during arthroscopy (menisci, ligaments, osteochondral defects);
* associated extraarticular lesions confirmed by magnetic resonance imaging (ligaments, tendons, bursae);
* lower limb axial deviation confirmed by whole leg weight-bearing radiograph; knee trauma in patients history;
* body mass index (BMI) higher than 35;
* hyaluronic acid intraarticular injection 6 months prior the arthroscopy and up to last follow-up control;
* steroids intraarticular injection 3 months prior the arthroscopy and up to last follow-up control;
* symptomatic slow acting drugs for osteoarthritis (SYSADOA) and/or non-steroidal anti-inflammatory drugs (NSAID) administration during the PRP treatment;
* systemic autoimmune rheumatic and/or polyarticular disease; gout, pseudogout and hyperuricaemia.
* Other exclusion criteria included: non-informed consent; treated knee injury during the PRP therapy; PRP injection cycle not completed; impediments to fill out the questionnaires; blood disease and/or immunosuppressant treatment and/or dicoumarol therapy; immunosuppressant and/or neoplastic and/or infectious diseases.

Ages: 31 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change of the width of cartilage in the knee joint assessed by magnetic resonance imaging before and after nine Platelets Rich Plasma injections. | 11 months after first Platelets Rich Plasma injection
  50 patients with Grade II or III chondromalatia in the knee joint, underwent one year treatment with autologous Platelets Rich Plasma. Magnetic resonance imaging was used to evaluate cartilage thickness and degree of degeneration before and after the treatement of nine Platelets Rich Plasma injection.

SECONDARY OUTCOMES:
Changes in the subjective and objective clinical outcomes before and after nine Platelets Rich Plasma injections. | 11 months
  50 patients with Grade II or III chondromalatia in the knee joint, underwent one year treatment with autologous Platelets Rich Plasma. To carefully assess the subjective and objective clinical outcomes, these questionnaires were used: Lysholm score, Tegner activity score, IKDC scores, and Cincinnati score. All these scores were recompleted 11 months after the beginning of the Platelets Rich Plasma injections.

CONTACTS AND LOCATIONS:
Overall Officials: Radek Hart, prof, M.D., Principal Investigator — Hospital Znojmo
Locations (1):
- Hospital Znojmo, Znojmo, Czechia

REFERENCES:
- See also: web site of Investigator´s institution — http://nemzn.cz